CLINICAL TRIAL: NCT04032535
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of CHF 6523 After Single or Multiple Ascending Doses in Healthy Subjects, Followed by a Placebo Controlled Repeated Dose 2-way Crossover in COPD Subjects
Brief Title: Investigate the Safety, Tolerability and Pharmacokinetics of CHF6523 in Healthy and in COPD Subjects
Acronym: CHF6523
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-06523AA1-01; 2018-004162-34 (EudraCT Number)
Record Dates: First submitted 2019-07-17; First posted 2019-07-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: COPD
Keywords: anti-inflamatory; PI3K; Sputum; COPD; inhaled
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: SAD and MAD in healthy volunteers plus 2way crossover in COPD patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SAD (Experimental): Single Ascending Dose of 2 cohorts:
  Cohort A will be administered three ascending dose levels: 0.2 mg (dose 1), 2 mg (anticipated dose 3), 8 mg (anticipated dose 5) or placebo; Cohort B will be administered three ascending dose levels: 1 mg (anticipated dose 2), 4 mg (anticipated dose 4), 14 mg (anticipated dose 6, maximum dose) or placebo.
  Interventions: Drug: CHF6523
- MAD (Experimental): Multiple Ascending Dose of 4 cohorts:
  Cohort A will be administered with 2 mg (anticipated dose 1) or placebo; Cohort B will be administered with 4 mg (anticipated dose 2) or placebo; Cohort C will be administered with 8 mg (anticipated dose 3) or placebo; Cohort D will be administered with 12 mg (anticipated dose 4) or placebo;
  Interventions: Drug: CHF6523
- 2way crossover (Experimental): Two 28-day treatment periods (Period 1 and Period 2), separated each by 32 days (up to 40 days) wash-out period, in crossover design. The treatment period will consist in repeated administrations of CHF 6523 at one dose level or placebo.
  Interventions: Drug: CHF6523

INTERVENTIONS:
Drug: CHF6523 — CHF6523 is a PI3K inhibitor (phosphoinositide3-kinase)

SUMMARY:
This study is designed to investigate the safety, tolerability and pharmacokinetics of inhaled CHF6523 DPI in healthy male subjects first and then in COPD subjects after single or repeated dosesof CHF6523. As an exploratory assessment, the anti-inflammatory effect of CHF6523 in COPDsubjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedures;
2. Male and female aged ≥40 years;
3. A female is eligible to enter the study if she is of non-childbearing potential i.e.

   physiologically incapable of becoming pregnant (e.g. postmenopausal women defined as being amenorrheic for ≥12 consecutive months without an alternative medical cause. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels, according to local laboratory ranges) or women permanently sterilized (e.g. bilateral oophorectomy, hysterectomy or bilateral salpingectomy or non-fertile partner). Women physiologically capable of becoming pregnant [i.e. women of childbearing potential (WOCBP)] are eligible to enter the study if they have negative pregnancy test at screening and are fulfilling one of the following criteria:
   1. WOCBP with fertile male partners;
   2. WOCBP with non-fertile male partners;
4. Male fulfilling one of the following criteria:

   1. Male with non-pregnant WOCBP partners;
   2. Male with pregnant WOCBP partner;
5. Subject with an established diagnosis of COPD (according to GOLD guidelines, update 2019 [7]) at least 12 months prior to the screening visit;
6. Subject with a smoking history of at least 10 pack-years [pack-years=number of cigarettes per day x number of years/20]. Current and ex- smokers are eligible. (Smoking cessation must be at least 6 months prior to the screening. If the subjects undergo smoking cessation therapy, it must be completed 6 months prior to the screening visit);
7. Subject with a BMI in the range of 19-32 kg/m2 extremes included;
8. Subject with a post-bronchodilator FEV1 ≥30% and ≤70% of the subject normal predicted value and a post-bronchodilator FEV1/FVC ratio <0.70 measured 10-15 minutes after 400 μg (4 puffs x 100 μg) of salbutamol pMDI. If this criterion is not met at screening, the test could be repeated once prior to randomisation visit;
9. Subject with at least one COPD exacerbation [i.e. resulting in the use of systemic (oral/IV/IM) corticosteroids and/or antibiotics or visit to an emergency department or hospitalisation] in the 12 months preceding the screening visit;
10. Subject on maintenance dual therapy with LABA/LAMA fixed combination within at least 2 months prior to screening visit;
11. Subject with a history of chronic bronchitis defined as chronic cough and sputum production for more than three months per year for two or more years and known as 'spontaneous sputum producer' subject;
12. Subject must be able to produce an adequate induced sputum sample defined as a load of at least 300 mg with a viability factor of not less than 70% (with less than 30% epithelial cells) at screening. The subject may be re-challenged once, if the first sputum sample does not meet these criteria;
13. Subject must be symptomatic at screening defined as having a CAT score ≥18;
14. Subject must be able to be trained to correctly use the DPI inhalers and to generate sufficient PIF (at least 40 L/min) using the In-Check Dial device at screening and prior to randomisation;
15. Subject must have a cooperative attitude and ability to perform the required outcome measurements (e.g. spirometry testing, induced sputum...).

Exclusion Criteria:

1. Pregnant or lactating female subject;
2. Subject with a current diagnosis of asthma;
3. Subject who have received or are planned to receive any type of vaccination within 3 weeks of their first dose of investigational product;
4. Subject with a COPD exacerbation [i.e. resulting in the use of systemic (oral/IV/IM) corticosteroids and/or antibiotics or visit to an emergency department or hospitalisation] or a lower respiratory tract infection within 6 weeks prior to screening visit or between screening and randomisation;
5. Subject on any maintenance therapy other than LABA/LAMA fixed combination within 2 months prior to screening visit;
6. Subject receiving treatment with one or more drugs, and related time windows, listed in the prohibited medication section (see section 5.2.2);
7. Subject requiring long-term (at least 12 hours daily) oxygen therapy for chronic hypoxemia;
8. Subject participating to a pulmonary rehabilitation programme or completing such a programme within the last 6 weeks prior to screening visit;
9. Subject with known respiratory disorders other than COPD that in investigator's opinion would affect efficacy and safety evaluation or place the subject at risk.

   This can include but is not limited to known -1 antitrypsin deficiency, active tuberculosis, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease;
10. Subject having lung cancer or a history of lung cancer;
11. Subject with active cancer or a history of cancer (other than lung) with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases). Localized carcinoma e.g. basal cell carcinoma (without metastases), in situ carcinoma of the cervix adequately treated is acceptable;
12. Subject with a known history of intolerance/hypersensitivity to any of the excipients/components contained in any of the formulations used in the trial;
13. Subject with a diagnosis of depression associated with suicidal ideation or behavior or with a diagnosis of generalised anxiety disorder that in the investigator's opinion would place the subject at risk;
14. Subject who has known history of clinically significant cardiovascular conditions such as, but not limited to, unstable or acute ischemic heart disease within one year prior to screening visit, NYHA Class III/IV heart failure, known history of sustained and non-sustained cardiac arrhythmias or history of atrial fibrillation diagnosed in the last 6 months prior to screening visit and not controlled with therapy rate control strategy;
15. Subject who has clinically significant abnormal 12-lead ECG that, in the investigator's opinion, would affect safety, PK or PD evaluation or place the subject at risk at screening or at randomisation visits;
16. Male subject with a QTcF >450 ms and female subject with a QTcF >470 ms at screening or at randomisation visits;
17. Subject with a history or symptoms of significant neurological disease including transient ischemic attack (TIA), stroke, seizure disorder or behavioural disturbances;
18. Subject who has unstable concurrent disease: e.g. uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; significant hepatic impairment, significant renal impairment; history of cerebrovascular disease; uncontrolled gastrointestinal disease (e.g. active peptic ulcer, Crohn's disease, ulcerative colitis, enteritis, unexplained diarrhea, bloody or loose stools); uncontrolled haematological disease; uncontrolled autoimmune disorders (e.g. rheumatoid arthritis, inflammatory bowel disease) or other disease or condition.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | Up to 4 weeks
  The number of events and the number and percentage of subjects experiencing TEAEs, treatment emergent ADRs, serious TEAEs, non-serious TEAEs, severe TEAEs, TEAEs leading to discontinuation of study drug and TEAEs leading to death will be presented by treatment.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC0-24h, | On Day 1 at pre-dose,10, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose.
  Dose proportionality of CHF 6523 for AUC0-24h, and classical PK parameters will be calculated
Cardiac Safety | At screening visit and on Day 1 at pre-dose, 10, 15, 30, 45 minutes and 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose and at 24 hours post dose;
  ECG QT Interval: Through digitised 12-lead ECG Extracted from 12-Lead 24h Holter ECG

OTHER OUTCOMES:
Concentration of sputum biomarkers in COPD patients | On Day 1 at pre-dose and on Day 28 after the dose
  Target Biomarkers in sputum supernatant, IL-6: change from baseline to end of treatment (mean of Day 24 and Day 28 values)
Concentration of blood biomarkers in COPD patients | On Day 1 at pre-dose and on Day 28 after the dose
  Target Biomarkers in plasma, IL-6, as change from baseline to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Govoni M, Bassi M, Girardello L, Lucci G, Rony F, Charretier R, Galkin D, Faietti ML, Pioselli B, Modafferi G, Benfeitas R, Bonatti M, Miglietta D, Clark J, Pedersen F, Kirsten AM, Beeh KM, Kornmann O, Korn S, Ludwig-Sengpiel A, Watz H. CHF6523 data suggest that the phosphoinositide 3-kinase delta isoform is not a suitable target for the management of COPD. Respir Res. 2024 Oct 19;25(1):380. doi: 10.1186/s12931-024-02999-5. PMID 39427187